CLINICAL TRIAL: NCT04418193
Title: Therapeutic Management in Patients With COVID-19 Infection at Risk of Secondary Aggravation: Patient Preference Trial Comparing Routine Care, Treatment With Hydroxychloroquine or Treatment With Hydroxychloroquine Plus Azithromycin
Brief Title: Patient Preference Trial for COVID-19 (PPT-COVID)
Acronym: PPT-COVID
Status: Withdrawn | Type: Observational
Why Stopped: treatments are no longer proposed to this type of patients
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 20-08
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date no treatment has proven its effectiveness in the caring of patients infected with type 2 Coronavirus. The Centre Hospitalier Princesse Grace (CHPG) has decided to only propose randomized double-blind placebo-controlled clinical trials to patients at the early and symptomatic stages of the disease. Data from the literature show in vitro results on the potential clinical benefit of some treatments such as chloroquine or hydroxychloroquine (HXCQ). Observational data suggest a potential benefit of this treatment alone or in combination with azithromycin (HXCQ + AZ). These data were advertised or led to a request from ambulatory medicine and patients to have access to these treatments despite their poor level of evidence. This leads to a decrease in the number of patients recruitable for clinical trials because they refuse the concept of control arms or they wish active treatment (CQ, HXCQ or HXCQ + AZ) from the start.

In this context, we propose to conduct in parallel with randomized trials, a so-called "patient preference" protocol which, after patients information, gives them the choice, either to participate in the trial or to choose between treatment with HXCQ, treatment with HXCQ + AZ or standard of care without medication. The patients follow-up and the main endpoint will be the same under the patient preference protocol as for the randomized trial.

The advantage of this approach is to offer a common follow-up to all patients, to take into account patients who refuse to participate in the clinical trial, to obtain external validity data, to reduce selection bias and to increase the heterogeneity of patients exposed to treatment options.

The expected objective is to see if the patient preference protocol leads to observe the same effects as in the randomized trial.

DETAILED DESCRIPTION:
Conduct of the research

* Pre-selection / Recruitment It is proposed to participate in the study to patients who cannot or do not wish to participate in a randomized therapeutic trial.
* Inclusion procedure During the inclusion visit, if the patient meets the study selection criteria, the investigator delivers oral and written information and responds to any patient questions.
* Follow-up of people suitable for research

  1. Inclusion visit The treatment chosen by the patient is administered. Socio-demographic, history, clinical and biological data are collected.
  2. Visit on day 3 ± 1 Hydroxychloroquinemia is dosed.
  3. Visit on day 5 ± 1 A nasopharyngeal swab sample is collected during the routine visit. This sampling is only performed for patients for whom the diagnosis of COVID-19 has been made by RT-PCR.
  4. Visit on day 10 ± 1 A nasopharyngeal swab sample is collected during the routine visit. This sampling is only performed for patients for whom the diagnosis of COVID-19 has been made by RT-PCR. Hydroxychloroquinemia is dosed.
  5. Visit on day 14 A visit or a telephone call is made to gather the occurrence of clinical events of interest on day 14. The treatments received during the last 14 days are collected.
  6. Visit on day 28 A visit or a telephone call is made to gather the occurrence of clinical events of interest on day 28.

The treatments received during the last 14 days are collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+)
* Infection with COVID-19 diagnosed by positive RT-PCR SARS-CoV-2 or, if not performed, by thorax CT-scan suggesting viral pneumonia of peripheral predominance in a clinically significant context.
* Diagnosed within the previous 48 hours.
* Having at least one of the following two risk factors for complications:
* age ≥75 years old
* Peripheral oxygen saturation (SpO2) ≤ 94% while breathing ambient air, or a partial oxygen pressure (PaO2) to fraction of inspired oxygen (FiO2) ratio ≤ 300 mmHg.
* Patients affiliated with or benefitting from a social security scheme
* Written and signed consent of the patient or a relative or, if not possible, emergency inclusion procedure
* Electrocardiogram showing absence of QT prolongation greater than 440 ms in men and 460 ms in women.
* Patient that can't or don't want to participate to a randomized clinical trial

Exclusion Criteria:

* Age below 18-year of age
* Negative RT-PCR SARS-CoV-2
* Peripheral capillary oxygen saturation less than or equal to 94% (SpO2≤94%) despite oxygen therapy greater than or equal to 3 L/min (≥ 3 L/min)
* Organ failure requiring admission to a resuscitation or high dependency unit
* Comorbidity that is life-threatening in the short-term (life expectancy <3 months)
* Any reason that makes follow-up at day 28 impossible
* Current treatment with hydroxychloroquine or hydroxychloroquine plus azithromycin
* Absolute contraindication to treatment with hydroxychloroquine (known hypersensitivity, concomitant treatment with risk of torsades de pointe) or azithromycin (known hypersensitivity to azithromycin, erythromycin, other macrolide, ketolide, in association with rye ergot alkaloids, cisapride, colchicine or severe hepatic failure)
* glucose-6-phosphate dehydrogenase (G6PD) known deficit
* Porphyria
* Hypokaliemia < 3.5 mmol/L
* Electrocardiogram showing corrected QT prolongation greater than 440 ms in men and 460 ms in women
* Child C liver cirrhosis
* Chronic kidney failure with estimated glomerular filtration rate (GFR) ≤ 30 ml/min
* Pregnant, lactating or parturient women
* Patient included in a randomized clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with COVID-19 infection diagnosed by positive RT-PCR SARS-CoV-2 or, if not performed, by thorax CT-scan suggesting viral pneumonia of peripheral predominance in a clinically significant context that can't or don't want to participate to a randomized clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Number of death from any cause, or the need for intubation and mechanical ventilation during the 14 days following inclusion and start of treatment. | day 14
  Number of death from any cause, or the need for intubation and mechanical ventilation during the 14 days following inclusion and start of treatment.

SECONDARY OUTCOMES:
Number of death from any cause, or the need for intubation and mechanical ventilation during the 28 days following inclusion and start of treatment. | day 28
  Number of death from any cause, or the need for intubation and mechanical ventilation during the 28 days following inclusion and start of treatment.
Clinical evolution on the World Health Organisation (WHO) Ordinal Scale for Clinical Improvement (OSCI) for COVID-19 between day 0 and day 14 | day 14
  Clinical evolution on the World Health Organisation (WHO) Ordinal Scale for Clinical Improvement (OSCI) for COVID-19 between day 0 and day 14. Score is between 0 and 8, 8 being the worst.
Clinical evolution on the WHO Ordinal Scale for Clinical Improvement for COVID-19 between day 0 and day 28. | day 28
  Clinical evolution on the WHO Ordinal Scale for Clinical Improvement for COVID-19 between day 0 and day 28. Score is between 0 and 8, 8 being the worst.
Number of all-cause mortality at day 14 | day 14
  Number of all-cause mortality at day 14
Number of all-cause mortality at day 28 | day 28
  Number of all-cause mortality at day 28
Rate of positive severe acute respiratory syndrome (SARS)-coronavirus 2 (CoV-2) Reverse Transcriptase (RT) - Polymerase Chain Reaction (PCR) on nasopharyngeal samples at day 5 | day 5
  Rate of positive severe acute respiratory syndrome (SARS)-coronavirus 2 (CoV-2) Reverse Transcriptase (RT) - Polymerase Chain Reaction (PCR) on nasopharyngeal samples at day 5
Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal samples at day 10 | day 10
  Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal samples at day 10
The rate of venous thromboembolic events at day 28, documented and confirmed by an adjudication committee. | day 28
  The rate of venous thromboembolic events at day 28, documented and confirmed by an adjudication committee.
Number of all-cause mortality at day 28 in patients aged 75 and older | day 28
  Number of all-cause mortality at day 28 in patients aged 75 and older
Clinical evolution on the WHO OSCI scale for COVID-19 between day 0 and day 28 for patients aged 75 or older | day 28
  Clinical evolution on the WHO OSCI scale for COVID-19 between day 0 and day 28 for patients aged 75 or older. Score is between 0 and 8, 8 being the worst.
Rate of severe adverse events at day 28 | day 28
  Rate of severe adverse events at day 28
Number of all-cause mortality at day 14 in patients aged 75 and older | day 14
  Number of all-cause mortality at day 14 in patients aged 75 and older

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco